CLINICAL TRIAL: NCT00003613
Title: Phase I Trial of O6 Benzylguanine and BCNU in Cutaneous T-cell Lymphoma
Brief Title: O6-benzylguanine and Carmustine in Treating Patients With Stage IA-IIA Cutaneous T-cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03119; CWRU 6496; U01CA062502 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — O(6)-benzylguanine; Carmustine

ARMS (1):
- Treatment (O6-benzylguanine, carmustine) (Experimental): Patients receive O6-benzylguanine IV over 1 hour followed by topical carmustine once every 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: O6-benzylguanine; Drug: carmustine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: O6-benzylguanine — Given IV
  Other Names: BG
Drug: carmustine — Given topically
  Other Names: BCNU; BiCNU; bis-chloronitrosourea
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of carmustine given together with O(6)-benzylguanine in treating patients with stage I or stage II cutaneous T-cell lymphoma that has not responded to previous treatment. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the kinetics of AGT depletion in CTCL skin lesions. II. To determine the toxicity of low dose BCNU plus O6BG.

OUTLINE: This is a dose-escalation study of carmustine.

Patients receive O6-benzylguanine IV over 1 hour followed by topical carmustine once every 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of carmustine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CTCL, stages IA-IIA
* Performance status ECOG grade 0, 1, or 2
* Patients must have recovered from toxicity of prior treatment and have received no CTCL therapy other than emoliation for at least 4 weeks
* Patients must have signed a consent form indicating the investigational nature of the treatment and its potential side effects
* WBC > 4,000/ul
* ANC > 2,000/ul
* Platelets > 100,000/ul
* Bilirubin < 1.5 mg/dL
* SGOT within normal range
* Prothrombin time within normal range
* Creatinine =< 1.5 mg/dL or creatinine clearance >= 70 ml/min
* Calcium and electrolytes normal
* Glucose-controlled (diet and insulin) diabetes is permitted
* DLCO > 80% normal with the exception of patients who demonstrate clinically normal lung function based on history, physical examination, and chest x-ray as interpreted by the principal investigator
* Only those patients with biopsiable tumor and willing to undergo several biopsies will be eligible
* Must have failed 1 conventional treatment other than topical corticosteroids; this includes UVB, PUVA, topical mechlorethamine, electron beam, photopheresis, chemotherapy and immuno-modulatory agents such as cytokines

Exclusion Criteria:

* Patients with a prior treatment with a nitrosourea
* Patients with known central nervous system involvement or primary CNS malignancies will be ineligible
* Patients with performance status ECOG grade 3 or 4
* Pregnant women, women who are breast feeding infants, or women with reproductive potential not practicing adequate contraception, because of potential toxicity to the fetus or infant
* Patients with active infection
* Patients with pulmonary disease as determined by history, physical examination, chest X-ray or pulse oximetry
* CTCL patients with stage IIB-IVB disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1999-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Percent decrease of AGT in CTCL skin lesions, obtained from tissue samples | Baseline to 6 weeks
  Point and interval estimates of response using the binomial distribution will be obtained using data from patients with measurable or evaluable disease. If responses occur, then the mean and median duration of response will be determined. Statistical significance will be determined using the t test for analysis of continuous data.
MTD of carmustine estimated as the dose level which is one level below where >= 2 DLT are observed | 6 weeks
  Toxicities will be recorded and tabulated. Additional point and interval estimates for the MTD will be obtained using the methods of logistic regression of the proportion of patients experiencing a dose-limiting toxicity of grade >= 2 and by conventional regression of the mean dose-limiting toxicities on dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Apisarnthanarax N, Wood GS, Stevens SR, Carlson S, Chan DV, Liu L, Szabo SK, Fu P, Gilliam AC, Gerson SL, Remick SC, Cooper KD. Phase I clinical trial of O6-benzylguanine and topical carmustine in the treatment of cutaneous T-cell lymphoma, mycosis fungoides type. Arch Dermatol. 2012 May;148(5):613-20. doi: 10.1001/archdermatol.2011.2797. PMID 22250189